CLINICAL TRIAL: NCT02932722
Title: Effect of Propofol on Cardioprotective Role of Remote Ischemic Preconditioning (RIPC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yunseok Jeon, Principal Investigator, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RIPC_propofol; 1605-079-761 (Other: Seoul National University Hospital IRB)
Record Dates: First submitted 2016-09-26; First posted 2016-10-13 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Myocardial Infarction
Keywords: Propofol; Sevoflurane; Preconditioning
MeSH Terms: conditions — Myocardial Infarction | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Sham Comparator): Patients in the control group will be receive remote ischemic preconditioning before anesthetic induction (before exposure to any anesthetic).
  Interventions: Other: Control
- Propofol (Active Comparator): Patients in the propofol groups will be receive remote ischemic preconditioning after anesthetic induction using propofol, as a main anesthetic.
  Interventions: Drug: Propofol
- Sevoflurane (Active Comparator): Patients in the sevoflurane groups will be receive remote ischemic preconditioning after anesthetic induction using sevoflurane, as a main anesthetic.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Other: Control — Patients in the control groups do not receive any anesthetic during remote ischemic preconditioning.
  Other Names: Not receiving any anesthetic
  Arms: Control
Drug: Propofol — Patients in the propofol group receive propofol anesthesia during remote ischemic preconditioning.
  Other Names: Receiving propofol anesthesia
  Arms: Propofol
Drug: Sevoflurane — Patients in the sevoflurane group receive sevoflurane anesthesia during remote ischemic preconditioning.
  Other Names: Receiving sevoflurane anesthesia
  Arms: Sevoflurane

SUMMARY:
This study involves research using human subjects (cardiac surgical patients) to evaluate the effect of remote ischemic preconditioning (RIPC) on cardioprotective outcomes. RIPC applied to upper or lower extremities has been shown cardioprotective role by lowering release of cardiac troponin in patients with cardiac diseases. However, it is not clear whether anesthetics, such as propofol or sevoflurane, may impair the cardioprotective effect of RIPC in cardiac surgical patients. Therefore, the purpose of the study is to compare the effects of anesthetics on cardioprotection of RIPC in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
Patients undergoing cardiac surgery using cardiopulmonary bypass will be randomized to control, propofol, or sevoflurane group. Patients in the control group will receive remote ischemic preconditioning (RIPC) on their upper arms before anesthetic induction. Patients in the propofol or sevoflurane groups will receive RIPC after anesthetic induction using propofol or sevoflurane, respectively. In all patients, arterial blood samples will be obtained before and after each RIPC. From the samples, human dialysate will be obtained and perfused to rat heart through Langendorff apparatus before ischemia-reperfusion injury to the rat heart. Infarct size of the sectioned rat heart will be compared among the three - control, propofol, and sevoflurane - groups.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I~III patients undergoing cardiac surgery using cardiopulmonary bypass

Exclusion Criteria:

* Cardiac surgery without using cardiopulmonary bypass
* Descending thoracic aortic surgery
* Strenuous exercise, excessive alcohol or caffeine intake 24 hours before remote ischemic preconditioning
* Left ventricular ejection fraction < 30%
* Uncontrolled hypertension or diabetes mellitus
* Severe renal or hepatic dysfunction
* Patients on hemodialysis
* Patients with arterio-venous fistula on arms or any reason to protect arms
* Peripheral vascular or nerve disease, bleeding tendency
* Preoperative use of IABP, ECMO, or ventricular assist devices
* Emergency operation, redo operation
* Refuse to enroll
* Pregnancy
* Preoperative use of beta-blockers

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2018-02-07 (Actual); Study Completion 2018-02-07 (Actual)

PRIMARY OUTCOMES:
Infarct size of the rat heart | 1 day after ischemia-reperfusion injury

SECONDARY OUTCOMES:
Cardiac troponin I after surgery | 72 hours postoperatively
Major adverse cardiovascular and cerebrovascular events | Through study completion, average of 2 weeks before hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Yunseok Jeon, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No